CLINICAL TRIAL: NCT03612128
Title: The Effect of Upper Extremity Mirror Therapy on Cerebral Re-organization, Functional Motor Skills, Daily Life Activities and Health Related Quality of Life in Children With Spastic Hemiplegic Cerebral Palsy
Brief Title: The Effect of Mirror Therapy on Cerebral Re-organization, Functional Motor Skills, and Quality of Life in Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Korkem, Researcher, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7603
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Spastic Hemiplegic Cerebral Palsy
Keywords: cerebral palsy; mirror therapy; cerebral re-organization; upper extremity; daily life activities; functional motor capacity; motor functions
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups; Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: In this type of controlled clinical trials, the same subjects are used as experimental and control groups, ie both the new treatment method and the classical method or the placebo method are applied to the same subjects. The efficacy is applied to the new treatment method and on the other hand the classical method is applied on the same subjects at different times and the results are compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Children continued their traditional physiotherapy
  Interventions: Other: control group
- intervention group (Active Comparator): We applied mirror therapy in addition to traditional physiotherapy
  Interventions: Other: intervention group

INTERVENTIONS:
Other: control group — Children continued their traditional physiotherapy including upper limb exercises in three times a week for 8 week.
  Other Names: traditional physiotherapy
  Arms: control group
Other: intervention group — Participants allocated to the experimental group completed three times a week, 8-week mirror therapy in addition to traditional physiotherapy . This protocol consisted of mirror therapy with a mirror box.
  Other Names: mirror therapy in addition to traditional physiotherapy
  Arms: intervention group

SUMMARY:
The purpose of this study is to investigate brain reorganization, functional motor development, level of daily living activity and quality of life of upper extremity mirror therapy in children with spastic hemiplegic cerebral palsy. Several studies have reported increased use of the affected arm following rearrangement of cerebral re-organization with mirror therapy. The investigator's study is the first of its kind and was planned to evaluate the effectiveness of upper extremity mirror therapy in cerebral reorganization and functional motor skills in children with spastic hemiplegic cerebral palsy. Hypothesis of this study is that mirror therapy improves brain re-organisation, functional motor skills and daily living activities in unilateral spastic CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common neurodisability in children. It has been defined as a disorder of movement and posture due to a defect or lesion of the immature brain and as a group of non-progressive, but often changing motor impairment syndromes secondary to lesions or anomalies of the brain arising in the early stages of development.

Characteristically, children with unilateral cerebral palsy (CP) have one well-functioning hand and one impaired hand.Common features of the hemiplegic hand are slowness, abnormal muscle tone, decreased strength, and coordination difficulties, which occur to a varying extent in children independently of age. Many children also have impaired sensibility and mirror movements. Perhaps most importantly, children with unilateral CP hav e varying degrees of limitation in their ability to handle objects in daily life. This limitation is most obvious insituations where two hands are needed. However, knowledge about bimanual ability in chil dren with unilateral CP and its development over time is scarce at present.

To improve upper extremity function in children with unilateral CP, the mirror therapy is a promising approach. Mirror therapy for the first time, Ramachandran et al. has described for the treatment of phantom pain in amputee. Also in unilateral spastic CP mirror therapy have indicated that visual illusion of functional limb provided by mirror can support healing. By means of visual feedback, modified vision and perception is stimulated plasticity the premotor cortex and developed re-organization. In the current studies, mirror therapy in hemiplegic patients, have been shown that improve the function and reduce the sensitivity of the hemi neglect. Gygax et al. have investigated the effects of mirror therapy on upper extremity function 10 children with unilateral spastic CP between 6-14 years. Consequently, the spontaneous use affected hand, the maximum grip force increase of 15% and is demonstrated that improve the upper extremity motor function.

ELIGIBILITY:
Inclusion Criteria:

* Congenital spastic hemiplegic cerebral palsy,
* Between the ages of 4-18,
* Continuing physiotherapy and rehabilitation program throughout the study.

Exclusion Criteria:

* Upper extremity fracture or muscle-tendon and bone operation shortly before 6 months,
* Any pharmacologic agent that will inhibit spasticity within 6 months,
* Visual function disorder except eye fracture defect

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) | change from baseline brain reorganization at 8 weeks
  Brain reorganization was assessed by functional magnetic resonance imaging (fMRI).Being a non-invasive method, FMRI is nowadays the most common method used to map the neural activity of the human brain. fMRI is also used to describe patterns of cortical activation in children and adults with brain lesions
Quality of upper extremity skills assessment (QUEST) | change from baseline upper extremity skills at 8 weeks
  Quality of upper extremity skills assessment was be assessed by Quality of Upper Extremity Skills Test (QUEST). The test evaluates that handcraft and the quality of the movement in children with CP.This is an objective standardized measure evaluating the quality of upper extremity function in 4 domains: dissociated movement, grasp, protective extension, and weight bearing. Scores for the QUEST are calculated as percentages with a maximum score of 100.

SECONDARY OUTCOMES:
Functional independence measure (WeeFIM) | change from baseline functional independence at 8 weeks
  The functional independence assessment was be assessed by Functional Independence Measure (WeeFIM). The Weefim was designed as a basic indicator of severity of disability and to determine the amount of assistance required by children to perform daily living activities on a consistent basisThe subsets are categorized as self-care (six items), sphincter control (two items),transfers (three items), locomotion (two items), communication (two items), and social cognition (three items). Each measurement item of the subsets is scored on a scale of 1- 7, where 1 indicates total assistance and 7 shows complete independence. The minimum total score is 18 (total dependence in all skills) and the maximum score is 126 (complete independence in all skills).
Child Health Questionnaire Parent Form 50 Questions (CHQ-PF50) | change from baseline quality of life at 8 weeks
  Health related quality of life was evaluated by the Child Health Questionnaire Parent Form 50 Questions (CHQ-PF50). 50-item parent-completed CHQ (CHQ-PF50), which measures 11 domains of health. Physical domains include the following: physical functioning, role/social limitations as a result of physicalhealth, bodily pain/discomfort, and general health perception.
  Psychosocial domains include the following: role/social limitations as a result of emotional-behavioral problems, self-esteem, mental health, general behavior, emotional impact on parent, and time impact on parents. A separate domain measures limitations in family activities. There is also a single-item measure of family cohesion. Scores for the domains and single item range from 0 to 100, with higher scores indicating better HRQL

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Korkem, PhD, Study Director — Uskudar University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fedrizzi E, Pagliano E, Andreucci E, Oleari G. Hand function in children with hemiplegic cerebral palsy: prospective follow-up and functional outcome in adolescence. Dev Med Child Neurol. 2003 Feb;45(2):85-91. PMID 12578233
- [Background] Siebes RC, Wijnroks L, Vermeer A. Qualitative analysis of therapeutic motor intervention programmes for children with cerebral palsy: an update. Dev Med Child Neurol. 2002 Sep;44(9):593-603. doi: 10.1017/s0012162201002638. PMID 12227614
- [Background] Odding E, Roebroeck ME, Stam HJ. The epidemiology of cerebral palsy: incidence, impairments and risk factors. Disabil Rehabil. 2006 Feb 28;28(4):183-91. doi: 10.1080/09638280500158422. PMID 16467053
- [Background] Skold A, Josephsson S, Eliasson AC. Performing bimanual activities: the experiences of young persons with hemiplegic cerebral palsy. Am J Occup Ther. 2004 Jul-Aug;58(4):416-25. doi: 10.5014/ajot.58.4.416. PMID 15315248
- [Background] Gygax MJ, Schneider P, Newman CJ. Mirror therapy in children with hemiplegia: a pilot study. Dev Med Child Neurol. 2011 May;53(5):473-6. doi: 10.1111/j.1469-8749.2011.03924.x. Epub 2011 Mar 17. PMID 21410693